CLINICAL TRIAL: NCT00249145
Title: Risperidone in the Treatment of Behavioral Disturbances in Demented Patients: an International, Multicenter, Placebo-controlled, Double-blind, Parallel-group Trial Using Haloperidol as Internal Reference
Brief Title: A Study of the Effectiveness and Safety of Risperidone in the Treatment of Behavioral Disturbances in Patients With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006046
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular
Keywords: Dementia; Alzheimer's Disease; vascular dementia; mixed dementia, risperidone; nursing home
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Mixed Dementias | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to compare the safety and efficacy of risperidone (an antipsychotic medication) to that of placebo in the treatment of behavioral disturbances associated with dementia.

DETAILED DESCRIPTION:
Dementia is a term used for a collection of symptoms that can be caused by a number of diseases or injuries that affect the brain. Individuals with dementia have a loss of function in cognition (thinking, perception, learning, verbal communication, memory, judgment), which may lead to behavioral and personality changes (for example, agitation, delusions, hallucinations). Some causes of dementia are reversible; however, irreversible dementia is caused by certain conditions, such as Alzheimer's disease. Dementia is common in elderly individuals, but it is not a normal part of aging. This is a randomized, double-blind, parallel-group, placebo-controlled study comparing the effectiveness and safety of risperidone to placebo in patients with behavioral disturbances associated with dementia. Haloperidol is included as a reference therapy to confirm that the efficacy analyses are valid. The study is composed of two periods: a 1-week run-in period in which patients are discontinued from other antipsychotic drugs and take placebo twice daily and a 12-week double-blind treatment period. At the end of the run-in period, patients are randomly assigned to one of three risperidone doses, or placebo, or haloperidol (all oral solutions). The starting dose of risperidone and haloperidol is 0.25 milligrams (mg) twice daily, which is increased gradually to a maximum dose of 2 mg/day. If the patient does not have a sufficient response, the dose can be gradually increased to a maximum of 4 mg/day. The patient receives these doses for the remainder of the double-blind period. The primary measure of effectiveness is a reduction of >= 30% from baseline to the end of double-blind treatment on the total Behavior Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) score. The BEHAVE-AD is a rating scale used to evaluate behavior symptoms in patients with Alzheimer's disease. Additional efficacy measures include the Clinical Global Impressions (CGI), a rating system used to evaluate the overall and severity of clinical change in a patient with various diseases affecting the brain; the Cohen-Mansfield Agitation Inventory (CMAI), a questionnaire evaluating agitation; the Functional Assessment Staging (FAST), a diagnostic tool for determining the stage of dementia; and the Mini-Mental State Examination (MMSE), a clinical measure used to evaluate cognition. Safety evaluations include the incidence of adverse events; results of clinical laboratory tests (hematology, biochemistry, urinalysis); measurements of vital signs; physical and neurological examinations and electrocardiogram (ECG) findings; evaluations of the presence and severity of sedation; a computed tomography (CT) scan of the brain; and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone is more effective than placebo, as measured by a change from baseline on the total BEHAVE-AD score, in treating behavioral disturbances in demented patients. Risperidone oral solution 1 mg/mL; haloperidol oral solution, 1 mg/mL; placebo oral solution. Starting doses of 0.25 mg twice daily and increasing to 2 mg/day. If 2 mg/day shows an insufficient response, a maximum of 4 mg/day of risperidone or haloperidol is permitted. Total treatment duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dementia of the Alzheimer's type, mixed dementia, or vascular dementia, (as classified by the Diagnostic and Statistical Manual of Mental Diseases, 4th edition [DSM-IV]) and have behavioral disturbances
* a score >=4 on the FAST
* a score <=23 on the MMSE
* a BEHAVE-AD total score >=8, and a BEHAVE-AD global rating >=1
* must be institutionalized.

Exclusion Criteria:

* Patients with other medical or neurological conditions in which cognition (thinking, perception, learning, verbal communication, memory, judgment) is diminished (for example, drug overdosage, severe liver, heart, lung, and kidney malfunctions, Parkinson's disease)
* other psychiatric disorders, including major depression, schizophrenia, substance abuse or dependence
* abnormal electrocardiogram (ECG) findings
* abnormal clinical laboratory test findings.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 1995-04; Study Completion 1996-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of double-blind treatment on the total BEHAVE-AD score.

SECONDARY OUTCOMES:
Change from baseline to end of double-blind treatment in global rating, total BEHAVE-AD score, total CMAI score, CGI severity, FAST, and MMSE; safety evaluations conducted throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] De Deyn PP, Rabheru K, Rasmussen A, Bocksberger JP, Dautzenberg PL, Eriksson S, Lawlor BA. A randomized trial of risperidone, placebo, and haloperidol for behavioral symptoms of dementia. Neurology. 1999 Sep 22;53(5):946-55. doi: 10.1212/wnl.53.5.946. PMID 10496251
- [Derived] Roughley M, Mena C, Howard R, Reeves S, Bertrand J. Guiding safer risperidone prescribing in Alzheimer's disease with therapeutic drug monitoring. Br J Clin Pharmacol. 2023 Jul;89(7):2316-2321. doi: 10.1111/bcp.15692. Epub 2023 Feb 28. PMID 36791792